CLINICAL TRIAL: NCT03074773
Title: Paravertebral Block in Coarctation of the Aorta
Brief Title: The Effect of Paravertebral Block With Dexamethasone on Intraoperative and Postoperative Analgesia in Children Undergoing Surgery for Coarctation of Aorta
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Hassan Saleh, Lecture of anethesia, Cairo university, Cairo University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: N-81-2016
Record Dates: First submitted 2017-02-24; First posted 2017-03-09 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Coarctation of Aorta
MeSH Terms: conditions — Aortic Coarctation | interventions — Dexamethasone; Calcium Dobesilate; Ultrasonography; Bupivacaine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- paravertebral block with bupivacaine (Active Comparator): this group will receive 0.5mg/kg bupivacaine 0.25% diluted with isotonic saline (total volume 15ml) paravertebral block ultrasound guided pre-emptively
  Interventions: Device: ultrasound; Procedure: paravertebral block; Drug: Bupivacaine; Other: isotonic saline
- paravertebral block with bupivacaine and dexamethasone (Active Comparator): this group will receive 0.5mg/kg bupivacaine 0.25% mixed to 0.1 mg/kg dexamethasone diluted with isotonic saline (total volume 15ml) paravertebral block ultrasound guided pre-emptively
  Interventions: Drug: Dexamethasone; Device: ultrasound; Procedure: paravertebral block; Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone is commonly used in the perioperative period to reduce postoperative nausea and vomiting. Additionally, it has been reported to have analgesic effects.
  The analgesic effect of epidural or perineural dexamethasone administration is not clear. Dexamethasone might have a local anesthetic effect on nerve by direct membrane action
  Other Names: decadron
  Arms: paravertebral block with bupivacaine and dexamethasone
Device: ultrasound — The growth of ultrasound technology and, with it, our ability to visualize the pleura and other structures in and around the paravertebral space has fueled a tremendous increased interest in performing thoracic paravertebral blocks. These blocks may be used for acute pain control, as an adjunct to general anesthesia for peri-operative pain control and, in some practices, as the primary anesthetic
Procedure: paravertebral block — paravertebral block is an effective analgesic technique used in various types of surgery, trauma and chronic pain. it decreases postoperative pain and reduces opioid consumption which in turns improve postoperative pulmonary function hoping for early extubation.
Drug: Bupivacaine — it is an amino amide local anesthetic drug
  Other Names: marcain
Other: isotonic saline — sterile sodium chloride solution at physiological concentration (0.87%); used as diluting agent when added to local anesthetic drug
  Other Names: normal saline
  Arms: paravertebral block with bupivacaine

SUMMARY:
Anesthetic management for surgery of aortic coarctation needs special care due to severe pain during lateral thoracotomy incision, the intraoperative hemodynamic instability related to skin incision at lateral thoracotomy, clamping and declamping of the aorta, needs of large doses of analgesia perioperative, needs of vasodilators. Also, postoperative care of the patients after repair is very important issue. The investigators will compare the effect of para-vertebral block with bupivacaine alone or with dexamethasone on Intra and postoperative analgesia.

DETAILED DESCRIPTION:
The patients will be divided randomly by sealed envelope into 2 equal groups. Group I (n=30) will receive paravertebral block with 0.5mg/kg bupivacaine 0.25% diluted with isotonic saline (total volume 15ml) and group II (n=30) will receive paravertebral block with 0.5mg/kg 0.25% bupivacaine and 0.1mg/kg dexamethasone.intraoperative fentanyl needs, Intra and postoperative hemodynamics and OPS pain scores will be recorded. Possible risks as hypertension will be treated by nitroglycerin infusion 0.5ug/kg/min or tachycardia (HR more than 20% than baseline) will be managed by additional doses of fentanyl 1-2ug/kg, bradycardia (20% decrease from the baseline) will be managed by atropine 0.02mg/kg. Also, the complications of paravertebral block as peridural and intravascular injection can be avoided by careful aspiration before injection and injection while visualization of the needle by U/S.

ELIGIBILITY:
Inclusion Criteria:

* 4m-6 years males and females scheduled for surgery for coarctation of the aorta

Exclusion Criteria:

* patients with associated other cardiac anomalies (e.g. VSD), patients with airway abnormality, patients with heart failure, patients with endocrine disorders, patients with history of convulsions, neurological disorder, hepatic, renal and neuromuscular diseases, coagulopathy, history of hyperthermia, infection at site of the block and family history of hypersensitivity

Ages: 4 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-10-30 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Intraoperative fentanyl needs | 3hours
  total fentanyl consumption intraoperatively
postoperative analgesic requirements | 24hours
  total narcotic consumption

SECONDARY OUTCOMES:
the first time the analgesic required | 24 hours
  the time of narcotics need
extubation time | 24 hours
  postoperative extubation

CONTACTS AND LOCATIONS:
Overall Officials: kasr alaini hospital, Study Director — Cairo University
Locations (1):
- Amany Hassan Saleh, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saleh AH, Hassan PF, Elayashy M, Hamza HM, Abdelhamid MH, Madkour MA, Tawadros PZ, Omar H, Kamel MM, Zayed M, Helmy M. Role of dexamethasone in the para-vertebral block for pediatric patients undergoing aortic coarctation repair. randomized, double-blinded controlled study. BMC Anesthesiol. 2018 Nov 30;18(1):178. doi: 10.1186/s12871-018-0637-y. PMID 30501611